CLINICAL TRIAL: NCT00633139
Title: A Single Center, Open-Label, Non-Randomized, Uncontrolled, Multiple-Dose, Dose Escalation Study of the Safety, Pharmacokinetics, Efficacy and Long Term Safety of HGT-1111 (Recombinant Human Arylsulfatase A [rhASA, Metazym]) for the Treatment of Patients With Late Infantile Metachromatic Leukodystrophy (MLD)
Brief Title: Long-term Metazym Treatment of Patients With Late Infantile Metachromatic Leukodystrophy (MLD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGT-MLD-048; 2007-006345-40 (EudraCT Number)
Record Dates: First submitted 2008-02-29; First posted 2008-03-11 (Estimated); Results first posted 2012-06-15 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Late Infantile Metachromatic Leukodystrophy
Keywords: Metazym; Late infantile; Metachromatic leukodystrophy; Long-term safety
MeSH Terms: conditions — Leukodystrophy, Metachromatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Cohort 1: 50 U/kg Recombinant human Arylsulfatase A (rhASA)
  Interventions: Biological: Recombinant human Arylsulfatase A (rhASA)
- Cohort 2 (Experimental): Cohort 2: 100 U/kg Recombinant human Arylsulfatase A (rhASA)
  Interventions: Biological: Recombinant human Arylsulfatase A (rhASA)
- Cohort 3 (Experimental): Cohort 3: 200 U/kg Recombinant human Arylsulfatase A (rhASA)
  Interventions: Biological: Recombinant human Arylsulfatase A (rhASA)

INTERVENTIONS:
Biological: Recombinant human Arylsulfatase A (rhASA) — intravenous infusion, every other week for 26 weeks
  Other Names: Metazym; HGT-1111

SUMMARY:
This is a single center, open-label study of patients with late infantile MLD. All patients were previous treated 26 weeks in the phase I trial (EudraCT number: 2006-005341-11, NCT00418561). All patients will be offered continuing treatment in this study and will in this protocol receive 13 infusions, whereby the patients total have had 27 infusions of Metazym. One infusion will be given every other week. After a total of 52 weeks of treatment the subjects will continue treatment in a compassionate use protocol. Safety (AE/SAE) will be monitored at every visit.

ELIGIBILITY:
Inclusion Criteria:

The patients from the Phase I trial must meet the following criteria to be enrolled in the study.

* Subject's legally authorized guardian(s) must provide signed, informed consent prior to performing any study-related activities (trial-related activities are any procedures that would not have been performed during normal management of the subject)
* The subject and his/her guardian(s) must have the ability to comply with the clinical protocol

Exclusion Criteria:

* Spasticity so severe to inhibit transportation
* Presence of known clinically significant cardiovascular, hepatic, pulmonary or renal disease or other medical condition that, in the opinion of the Investigator, would preclude participation in the trial
* Any other medical condition or serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the trial
* Use of any investigational product other than rhASA within 30 days prior to study enrolment or currently enrolled in another study which involves clinical investigations

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2007-01-22 (Actual); Primary Completion 2008-11-25 (Actual); Study Completion 2008-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- PhaseOneTrials A/S, Hvidovre, Denmark

REFERENCES:
- [Derived] I Dali C, Groeschel S, Moldovan M, Farah MH, Krageloh-Mann I, Wasilewski M, Li J, Barton N, Krarup C. Intravenous arylsulfatase A in metachromatic leukodystrophy: a phase 1/2 study. Ann Clin Transl Neurol. 2021 Jan;8(1):66-80. doi: 10.1002/acn3.51254. Epub 2020 Dec 17. PMID 33332761

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children with an established diagnosis of late metachromatic leukodystrophy (MLD) due to arylsulfatase A (ASA) deficiency were recruited.
Pre-assignment Details: All participants that completed study recombinant human arylsulfatase A (rhASA-01) (NCT00418561) except 1 participant who did not complete (at week 18) the rhASA-01 (NCT00418561) participated in HGT-MLD-048/rhASA-03 (NCT00633139).
Groups:
- Cohort 1: Participants received a single dose of rhASA at 25 units per kilogram (U/kg) intravenous (IV) infusion in rhASA-01 (NCT00418561) study. Thereafter a repeated dose of rhASA at 50 U/kg, over 30 minutes was administered every other week up to Week 52.
- Cohort 2: Participants received a repeated dose of rhASA at 100 U/kg IV infusion over 30 minutes was administered every other week up to Week 52.
- Cohort 3: Participants received a repeated dose of rhASA at 200 U/kg IV infusion over 60 minutes was administered every other week up to Week 52.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 4 | 5 | 4
Completed | 4 | 4 | 3
Not Completed | 0 | 1 | 1
Not completed — Non compliance | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Participants received a single dose of rhASA at 25 U/kg IV infusion in rhASA-01 (NCT00418561) study. Thereafter a repeated dose of rhASA at 50 U/kg, over 30 minutes was administered every other week up to Week 52.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 4 | 5 | 4 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 5 | 4 | 13
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 36.25 (9.32) | 41.80 (10.13) | 30.75 (7.27) | 36.69 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 8
  Male | 2 | 2 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 4 | 5 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Relative Changes (%) in Gross Motor Function Measurement (GMFM)
Description: Change (percent change) in GMFM is measured from baseline to end of study (Week 52). GMFM is measured using GMFM-88. The GMFM-88 item scores can be summed to calculate a total GMFM-88 score. For each GMFM-88 item, the score is between 0 (minimal) to 3 (maximum). The total GMFM-88 score is between 0 (minimal) to 264 (maximum). Relative changes in GMFM are calculated as percentage change from baseline divided by the age difference in months between first and last visit. The GMFM score decreases over time, which, indicates that the disease worsened over time. Score over time (SOT), data mentioned over mean represents the adjusted mean.
Time Frame: Baseline, 52 Weeks
Population: Intent to Treat (ITT) population included all the participants in the study.
Measure: Mean (95% Confidence Interval); unit: Relative % change in total GMFM-88 SOT
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
Relative % change in total GMFM-88 SOT | -2.98 [-6.08 to 0.12] | -5.42 [-8.50 to -2.34] | -5.28 [-8.91 to -1.65]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2 vs Cohort 3; Test type: Superiority or Other; p = 0.4013, ANCOVA

2. Primary Outcome: Relative Change in Mullen's Scales of Early Learning
Description: Changes in Mullen's Scales of Early Learning are measured from baseline to end of study (Week 52) using Mullen's Scales of Early Learning. T scores, percentile ranks, and age equivalents can be computed for the four scales separately (visual reception, fine motor, expressive language, and receptive language). Relative change is calculated as percentage change from baseline divided by the age-difference in months between first and last visit. When Mullen's score decreases over time, it indicates the disease worsened over time. Data mentioned over mean represents the adjusted mean.
Time Frame: Baseline, 52 Weeks
Population: ITT population.
Measure: Mean (95% Confidence Interval); unit: Relative % change in Mullen's SOT
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
Relative % change in Mullen's SOT | -2.82 [-6.31 to 0.66] | -2.97 [-6.47 to 0.54] | -6.98 [-11.95 to -2.01]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2 vs Cohort 3; Test type: Superiority or Other; p = 0.2750, ANCOVA

3. Secondary Outcome: Change in Cerebrospinal Fluid (CSF) Sulfatide
Description: Changes in CSF sulfatide from baseline to end of study (Week 52). Data mentioned over mean represents the adjusted mean.
Time Frame: Baseline, 52 Weeks
Population: ITT population
Measure: Mean (95% Confidence Interval); unit: %change in CSF sulfatide
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
%change in CSF sulfatide | 8.60 [-0.77 to 17.97] | -1.53 [-8.63 to 5.56] | -2.77 [-14.35 to 8.81]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2 vs Cohort 3; Test type: Superiority or Other; p = 0.1363, ANCOVA

ADVERSE EVENTS:
Time Frame: 52 weeks of treatment
Description: All other adverse events (AEs) (>5% reporting frequency) reported here are either probable (PRB) or definitely (DEF) related to drug administration.
Groups:
- Cohort 1: Cohort 1: Participants received a single dose of rhASA at 25 U/kg IV infusion in rhASA-01 (NCT00418561) study. Thereafter a repeated dose of rhASA at 50 U/kg, over 30 minutes was administered every other week up to Week 52.
- Cohort 2: Cohort 2: Participants received a repeated dose of rhASA at 100 U/kg IV infusion over 30 minutes was administered every other week up to Week 52.
- Cohort 3: Cohort 3: Participants received a repeated dose of rhASA at 200 U/kg IV infusion over 60 minutes was administered every other week up to Week 52.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Serious Adverse Events (participants affected / at risk) | 2/4 | 2/5 | 3/4
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=5) | Cohort 3 (N=4)
malnutrition (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (3)
bronchitis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
blindness (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
post procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
peritonitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=5) | Cohort 3 (N=4)
Feeding tube complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Medical device complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood iron decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood iron increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Drug specific antibody present (Investigations) | 2 (2) | 0 (0) | 0 (0)
General physical condition abnormal (Investigations) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Leukodystrophy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 2 (5) | 2 (3) | 1 (1)
Hypotonia (Nervous system disorders) | 2 (5) | 4 (5) | 3 (4)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle spasticity (Nervous system disorders) | 4 (6) | 4 (7) | 1 (1)
Mutism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Speech disorder developmental (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 2 (15) | 2 (16) | 3 (11)
Pyrexia (General disorders) | 3 (6) | 3 (4) | 3 (5)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Herpangina (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Postoperative infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No